CLINICAL TRIAL: NCT00419536
Title: A Phase IA/IB, Two Arm, Multi-center, Open-label, Dose Escalation Study of Oral LBH589 Alone and in Combination With IV Docetaxel and Oral Prednisone in Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Safety of LBH589 Alone and in Combination With Intravenous Docetaxel and Prednisone
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589A2105
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2010-04

CONDITIONS: Hormone Refractory Prostate Cancer Disease
Keywords: LBH; LBH589; Prostate Cancer; HRPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Panobinostat

INTERVENTIONS:
Drug: LBH589

SUMMARY:
This 2-arm study is designed to determine the maximum tolerated dose of LBH589 as a single agent and in combination with docetaxel and prednisone 5 mg twice daily (second arm) and to characterize the safety, tolerability, biologic activity and pharmacokinetic profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hormone refractory prostate cancer
* Patients must have metastatic disease with at least 1 measurable soft tissue lesion that can be assessed by CT or MRI and/or detectable lesion(s) on bone scintigraphy scan. Patients with only elevated PSA levels are not eligible for entry.
* Patients must meet laboratory inclusion criteria defined in the protocol
* Patients must be able to provide written informed consent

Exclusion Criteria:

* Patients with prior or concurrent brain metastases
* Impaired cardiac, gastrointestinal, kidney or liver function
* Use of therapeutic androgens Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108
Dates: Start 2006-05

PRIMARY OUTCOMES:
To determine the maximum tolerated dose

SECONDARY OUTCOMES:
Safety
Tolerability
Biologic activity
Pharmacokinetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York